CLINICAL TRIAL: NCT07343830
Title: The Role of Preoperative Inflammation Markers, Renal Function, and Perfusion Stress in Predicting Acute Kidney Injury After Cardiac Surgery Under Cardiopulmonary Bypass: A Retrospective Cohort Study
Brief Title: Prediction of Acute Kidney Injury After Cardiac Surgery With Cardiopulmonary Bypass
Acronym: AKI-CPB
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet Akif Yilmaz, Principal Investigator, Ataturk University
Other Study IDs: AKI-CPB-RETRO-2025; 2026/1 (Other: Atatürk University Clinical Research Ethics Committee)
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Kidney Injury; Cardiac Surgery; Cardiopulmonary Bypass Surgery; Cardiac Surgery Associated - Acute Kidney Injury
Keywords: Acute kidney injury; Cardiac surgery; Cardiopulmonary bypass; Inflammatory markers; Neutrophil to lymphocyte ratio; Systemic immune inflammation index; C-reactive protein albumin ratio; Renal perfusion; Perfusion stress; KDIGO
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative AKI: Patients who developed acute kidney injury within 72 hours after cardiac surgery under cardiopulmonary bypass, defined according to the KDIGO serum creatinine criteria.
- No Postoperative AKI: Patients who did not develop acute kidney injury within 72 hours after cardiac surgery under cardiopulmonary bypass according to the KDIGO serum creatinine criteria.

SUMMARY:
Acute kidney injury (AKI) is a common and serious complication following cardiac surgery performed under cardiopulmonary bypass and is associated with increased morbidity, mortality, and prolonged hospital stay. Despite advances in perioperative management, the ability to accurately predict postoperative AKI remains limited.

Recent evidence suggests that preoperative inflammatory markers derived from routine laboratory tests, as well as indicators of intraoperative perfusion stress, may play an important role in the development of AKI. However, data evaluating these factors together in patients undergoing cardiac surgery with cardiopulmonary bypass are limited.

This retrospective observational cohort study aims to investigate the association between preoperative renal function, inflammatory indices, and intraoperative perfusion-related parameters with the development of postoperative AKI. Acute kidney injury will be defined according to the KDIGO serum creatinine criteria within the first 72 hours after surgery. The findings of this study may help identify patients at increased risk for AKI and contribute to improved perioperative risk stratification in cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a frequent complication after cardiac surgery performed under cardiopulmonary bypass (CPB) and represents a major determinant of short- and long-term adverse outcomes. The pathophysiology of postoperative AKI is multifactorial and involves hemodilution, non-pulsatile flow, ischemia-reperfusion injury, systemic inflammatory response, and alterations in renal perfusion during CPB. Despite similar surgical and anesthetic management, not all patients develop AKI, suggesting that preoperative patient-related factors and intraoperative perfusion stress play a critical role.

In recent years, easily accessible inflammatory indices derived from routine hematological and biochemical parameters, such as the neutrophil-to-lymphocyte ratio, systemic immune-inflammation index, and C-reactive protein to albumin ratio, have been proposed as potential predictors of postoperative complications, including AKI. In addition, intraoperative parameters reflecting perfusion stress, such as cardiopulmonary bypass duration, arterial lactate levels, and acid-base disturbances, may further contribute to renal injury. However, studies evaluating these factors together in the setting of cardiac surgery with CPB are limited.

This single-center, retrospective observational cohort study will include adult patients who underwent cardiac surgery under cardiopulmonary bypass. Demographic data, comorbidities, preoperative laboratory parameters, echocardiographic findings, and intraoperative CPB-related variables will be collected retrospectively from institutional medical records. Acute kidney injury will be defined and staged according to the KDIGO serum creatinine criteria within 48-72 hours after surgery. Urine output criteria will not be evaluated due to limitations inherent to retrospective data collection.

The primary objective of the study is to identify independent predictors of postoperative AKI by assessing the combined effects of preoperative renal function, inflammatory markers, and intraoperative perfusion stress parameters. Secondary objectives include evaluation of AKI severity and in-hospital mortality. Multivariable logistic regression and receiver operating characteristic analyses will be used to determine the predictive value of selected parameters.

By improving understanding of the factors associated with postoperative AKI, this study aims to support better perioperative risk stratification and inform future prospective investigations in patients undergoing cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Patients who underwent cardiac surgery under cardiopulmonary bypass
* Coronary artery bypass grafting, valve surgery, or combined cardiac surgery
* Elective or emergency procedures

Exclusion Criteria:

* Preoperative end-stage renal disease requiring dialysis
* Preoperative serum creatinine level greater than 4.0 mg/dL
* Off-pump cardiac surgery
* Missing preoperative or postoperative serum creatinine data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery with cardiopulmonary bypass at a single tertiary care center.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Acute Kidney Injury | Within 72 hours after cardiac surgery
  Development of acute kidney injury within 72 hours after cardiac surgery performed under cardiopulmonary bypass. Acute kidney injury will be defined according to the KDIGO serum creatinine criteria, based on an increase in serum creatinine of ≥0.3 mg/dL within 48 hours or ≥1.5 times baseline within 7 days. Urine output criteria will not be evaluated due to the retrospective nature of the study.

SECONDARY OUTCOMES:
Severity of postoperative AKI (KDIGO stage) | Within 72 hours after cardiac surgery (postoperative days 0-3); assessed using the highest serum creatinine value measured every 12 hours (6 measurements)
  AKI severity will be classified as KDIGO Stage 1-3 based on the change between preoperative creatinine (measured within 48 hours preoperatively) and the highest postoperative serum creatinine within the first 72 hours
In-Hospital Mortality | From the date of cardiac surgery through hospital discharge (index hospitalization), assessed at hospital discharge (up to 90 days)
  All-cause mortality during the index hospitalization following cardiac surgery, determined from hospital records

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the retrospective nature of the study and institutional data protection and patient confidentiality regulations. Only de-identified aggregate data will be reported in publications.

REFERENCES:
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Lee JW, Sharma AR, Lee SS, Chun WJ, Kim HS. The C-reactive protein to albumin ratio predicts postoperative complication in patients who undergo gastrectomy for gastric cancer. Heliyon. 2020 Jun 15;6(6):e04220. doi: 10.1016/j.heliyon.2020.e04220. eCollection 2020 Jun. PMID 32577578
- [Background] Sun J, Qi Y, Wang W, Meng P, Han C, Chen B. Systemic Immune-Inflammation Index (SII) as a Predictor of Short-Term Mortality Risk in Sepsis-Associated Acute Kidney Injury: A Retrospective Cohort Study. Med Sci Monit. 2024 Jun 28;30:e943414. doi: 10.12659/MSM.943414. PMID 38937949
- [Background] Bi JB, Zhang J, Ren YF, Du ZQ, Wu Z, Lv Y, Wu RQ. Neutrophil-to-lymphocyte ratio predicts acute kidney injury occurrence after gastrointestinal and hepatobiliary surgery. World J Gastrointest Surg. 2020 Jul 27;12(7):326-335. doi: 10.4240/wjgs.v12.i7.326. PMID 32821341
- [Background] Huen SC, Parikh CR. Predicting acute kidney injury after cardiac surgery: a systematic review. Ann Thorac Surg. 2012 Jan;93(1):337-47. doi: 10.1016/j.athoracsur.2011.09.010. PMID 22186469
- [Background] Lannemyr L, Bragadottir G, Hjarpe A, Redfors B, Ricksten SE. Impact of Cardiopulmonary Bypass Flow on Renal Oxygenation in Patients Undergoing Cardiac Operations. Ann Thorac Surg. 2019 Feb;107(2):505-511. doi: 10.1016/j.athoracsur.2018.08.085. Epub 2018 Oct 23. PMID 30365961
- [Background] Lagny MG, Jouret F, Koch JN, Blaffart F, Donneau AF, Albert A, Roediger L, Krzesinski JM, Defraigne JO. Incidence and outcomes of acute kidney injury after cardiac surgery using either criteria of the RIFLE classification. BMC Nephrol. 2015 May 30;16:76. doi: 10.1186/s12882-015-0066-9. PMID 26025079
- [Background] Hobson CE, Yavas S, Segal MS, Schold JD, Tribble CG, Layon AJ, Bihorac A. Acute kidney injury is associated with increased long-term mortality after cardiothoracic surgery. Circulation. 2009 May 12;119(18):2444-53. doi: 10.1161/CIRCULATIONAHA.108.800011. Epub 2009 Apr 27. PMID 19398670